CLINICAL TRIAL: NCT00221091
Title: Clinical Study of Idiopathic Normal Pressure Hydrocephalus for Neurological Improvement
Brief Title: Study to Evaluate Efficacy of Shunt Operation for Idiopathic Normal Pressure Hydrocephalus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Translational Research Center for Medical Innovation, Kobe, Hyogo, Japan (Other)
Collaborators: Codman & Shurtleff (Industry); Johnson & Johnson (Industry); Nihon Medi-Physics Co., Ltd. (Industry); Daiichi Pharmaceuticals (Industry); Eisai Limited (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRI NPH 03-01
Record Dates: First submitted 2005-09-13; First posted 2005-09-22 (Estimated); Last update posted 2009-02-09 (Estimated); Status verified 2009-02

CONDITIONS: Idiopathic Normal Pressure Hydrocephalus
Keywords: idiopathic normal pressure hydrocephalus; shunt
MeSH Terms: interventions — Ventriculoperitoneal Shunt

INTERVENTIONS:
Procedure: ventriculo-peritoneal shunt

SUMMARY:
This study evaluates the efficacy of shunt operation for idiopathic normal pressure hydrocephalus, and determines the diagnostic value of noninvasive procedures commonly practiced in the clinic.

DETAILED DESCRIPTION:
Idiopathic normal pressure hydrocephalus (iNPH) is a syndrome characterized by ventricular dilatation due to disturbed cerebrospinal fluid (CSF) circulation, accompanied by gait disturbance, dementia and/or urinary incontinence without causative disorders. With the aging of Japanese society, the number of patients is increasing, requiring diagnostic and therapeutic guidelines for the improvement of the patients' quality of life and social care. Under such conditions, this project was made as the prospective study of iNPH on Neurological Improvement (SINPHONI ). This study aims 1) to establish methods for non-invasive diagnosis of iNPH, and 2) to demonstrate therapeutic outcome of shunting operation by Codman Hakim programmable valve (CHPV). In this protocol, the evaluation of validity on MRI, tap test, CT cisternography, and CBF (3D-SSP) will be done in the diagnosis, and manual of initial setting pressure in CHPV for prevention of overdrainage problems will be estimated by modified Rankin scale (as primary endpoint) and some another scales during 1 year.

ELIGIBILITY:
Inclusion Criteria:

Patients who had at least one more points of the triad (gait disturbance, cognitive impairment, and urinary incontinence) in Japan NPH grading scale revised, and had disproportionate ventriculomegaly (Evans index >0.3) with closing of the CSF space at high convexity on MRI. These patients must be diagnosed clinically other causative disorders, and ventricular dilatation due to disturbance of the cerebrospinal fluid (CSF) circulation. Be able to give informed consent.

Exclusion Criteria:

1) Cannot have an MRI scan 2) Has a problem with bleeding tendency and other serological examination. (liver enzyme and renal dysfunction, blood coagulopathy, and etc.) 3) Is unable to understand the risks of the testing and surgical therapy. 4) is tolerable for one year follow up after shunting operation.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110
Dates: Start 2004-09; Study Completion 2005-10

PRIMARY OUTCOMES:
modified Rankin scale

SECONDARY OUTCOMES:
cognitive function, NPH grading scale

CONTACTS AND LOCATIONS:
Overall Officials: Masatsune Ishikawa, M.D., Principal Investigator — Department of Neurosurgery, kitano Hospital, The Tazuke Kofukai Medical Research Institute. City: Osaka
Locations (1):
- Noto General Hospital, Nanao-shi, Ishikawa Pref., Japan

REFERENCES:
- [Derived] Nakajima M, Yamada S, Miyajima M, Kawamura K, Akiba C, Kazui H, Mori E, Ishikawa M; SINPHONI-2 Investigators. Tap Test Can Predict Cognitive Improvement in Patients With iNPH-Results From the Multicenter Prospective Studies SINPHONI-1 and -2. Front Neurol. 2021 Nov 2;12:769216. doi: 10.3389/fneur.2021.769216. eCollection 2021. PMID 34795635
- [Derived] Kameda M, Yamada S, Atsuchi M, Kimura T, Kazui H, Miyajima M, Mori E, Ishikawa M, Date I; SINPHONI and SINPHONI-2 Investigators. Cost-effectiveness analysis of shunt surgery for idiopathic normal pressure hydrocephalus based on the SINPHONI and SINPHONI-2 trials. Acta Neurochir (Wien). 2017 Jun;159(6):995-1003. doi: 10.1007/s00701-017-3115-2. Epub 2017 Mar 1. PMID 28251346
- [Derived] Ishikawa M, Hashimoto M, Mori E, Kuwana N, Kazui H. The value of the cerebrospinal fluid tap test for predicting shunt effectiveness in idiopathic normal pressure hydrocephalus. Fluids Barriers CNS. 2012 Jan 13;9(1):1. doi: 10.1186/2045-8118-9-1. PMID 22239832
- [Derived] Kawaguchi T, Hirata Y, Bundo M, Kondo T, Owaki H, Ito S, Hashimoto M, Ishikawa M. Role of computerized tomographic cisternography in idiopathic normal pressure hydrocephalus. Acta Neurochir (Wien). 2011 Oct;153(10):2041-8; discussion 2048. doi: 10.1007/s00701-011-1047-9. Epub 2011 May 25. PMID 21611722
- [Derived] Hashimoto M, Ishikawa M, Mori E, Kuwana N; Study of INPH on neurological improvement (SINPHONI). Diagnosis of idiopathic normal pressure hydrocephalus is supported by MRI-based scheme: a prospective cohort study. Cerebrospinal Fluid Res. 2010 Oct 31;7:18. doi: 10.1186/1743-8454-7-18. PMID 21040519
- See also: INPH(Idiopathic Normal Pressure Hydrocephalus)--only in Japanese — http://www.inph.jp/